CLINICAL TRIAL: NCT00635752
Title: Trauma-focused Cognitive-behavioural Therapy for Children: A Study of Process and Outcome.
Brief Title: Trauma-focused Cognitive-behavioural Therapy(TF-CBT) for Children: A Study of Process and Outcome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Collaborators: Norway: Directorate for Health and Social Affairs (Unknown)
Responsible Party: Principal Investigator, Tine K. Jensen, Professor, Norwegian Center for Violence and Traumatic Stress Studies
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: s-07442a(REK)
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: TF-CBT; Effectiveness study; Trauma; Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive trauma-focused cognitive behavioral therapy (TF-CBT)
  Interventions: Other: TF-CBT
- 2 (Active Comparator): Participants will receive sessions of treatment as usual (TAU)
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: TF-CBT — TF-CBT sessions will include trauma-focused treatment, and will teach participants behavioral and coping skills.
  Arms: 1
Other: Treatment as Usual (TAU) — Participants will receive regular therapy as is usually practiced in clinics
  Other Names: TAU
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Trauma focused cognitive behavioral therapy (TF-CBT)is more effective in the treatment of traumatized youth than treatment as usual(TAU).

DETAILED DESCRIPTION:
Children experiencing traumas, such as sexual abuse, physical abuse, domestic violence, serious accidents, or natural disasters, may develop severe health problems.

This study will examine the short and long-term effects of trauma-focused cognitive-behavioural therapy on children exposed to serious trauma, and moderating factors of treatment outcome.

The study will use a random control design, and will be implemented in regular clinical practice in Norway.

More knowledge within this field is important for practitioners as well as policy makers in planning interventions and therapy for children and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Children between the age of 10-18
* referred to a guidance clinic
* who have experienced trauma
* present with PTSD reactions
* participants and the primary caretaker must be able to speak Norwegian.

Exclusion Criteria:

* Severe psychosis
* Severe mental retardation.
* The youth must not have had severe conduct disorders previous to the trauma experience

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
PTSD | Before session, middle, end, one year follow-up, 18 month follow-up

SECONDARY OUTCOMES:
Parent distress | Before session, middle, end, one year follow-up, 18 month follow-up
Therapeutic alliance | After 1st. and 6th. session

CONTACTS AND LOCATIONS:
Overall Officials: Tine K Jensen, PhD, Principal Investigator — Norwegian Centre for Violence and Traumatic Stress Studies
Locations (1):
- Norwegian center for violence and traumatic stress studies, Oslo, Norway

REFERENCES:
- [Background] Holt T, Jensen TK, Wentzel-Larsen T. The change and the mediating role of parental emotional reactions and depression in the treatment of traumatized youth: results from a randomized controlled study. Child Adolesc Psychiatry Ment Health. 2014 Apr 8;8:11. doi: 10.1186/1753-2000-8-11. eCollection 2014. PMID 24712976
- [Background] Dittmann I, Jensen TK. Giving a voice to traumatized youth-experiences with Trauma-Focused Cognitive Behavioral Therapy. Child Abuse Negl. 2014 Jul;38(7):1221-30. doi: 10.1016/j.chiabu.2013.11.008. Epub 2013 Dec 22. PMID 24367942
- [Background] Ormhaug SM, Jensen TK, Wentzel-Larsen T, Shirk SR. The therapeutic alliance in treatment of traumatized youths: relation to outcome in a randomized clinical trial. J Consult Clin Psychol. 2014 Feb;82(1):52-64. doi: 10.1037/a0033884. Epub 2013 Jul 29. PMID 23895084
- [Background] Holt, T., Cohen, J. A., Mannarino, A., & Jensen, T. K. (2014). Parental Emotional Response to Children's Traumas. Journal of Aggression, Maltreatment & Trauma. 23(10), 1057-1071. doi: 10.1080/10926771.2014.953717
- [Result] Jensen TK, Holt T, Ormhaug SM, Egeland K, Granly L, Hoaas LC, Hukkelberg SS, Indregard T, Stormyren SD, Wentzel-Larsen T. A randomized effectiveness study comparing trauma-focused cognitive behavioral therapy with therapy as usual for youth. J Clin Child Adolesc Psychol. 2014;43(3):356-69. doi: 10.1080/15374416.2013.822307. Epub 2013 Aug 9. PMID 23931093
- [Result] Glad KA, Jensen TK, Holt T, Ormhaug SM. Exploring self-perceived growth in a clinical sample of severely traumatized youth. Child Abuse Negl. 2013 May;37(5):331-42. doi: 10.1016/j.chiabu.2013.02.007. Epub 2013 Mar 30. PMID 23548683
- [Result] Hukkelberg S, Ormhaug SM, Holt T, Wentzel-Larsen T, Jensen TK. Diagnostic utility of CPSS vs. CAPS-CA for assessing posttraumatic stress symptoms in children and adolescents. J Anxiety Disord. 2014 Jan;28(1):51-6. doi: 10.1016/j.janxdis.2013.11.001. Epub 2013 Dec 1. PMID 24361907
- [Derived] Ovenstad KS, Ormhaug SM, Jensen TK. The relationship between youth involvement, alliance and outcome in trauma-focused cognitive behavioral therapy. Psychother Res. 2023 Mar;33(3):316-327. doi: 10.1080/10503307.2022.2123719. Epub 2022 Sep 20. PMID 36125352
- [Derived] Ovenstad KS, Jensen TK, Ormhaug SM. Four perspectives on traumatized youths' therapeutic alliance: Correspondence and outcome predictions. Psychother Res. 2022 Jul;32(6):820-832. doi: 10.1080/10503307.2021.2011983. Epub 2021 Dec 10. PMID 34893017
- [Derived] Ovenstad KS, Ormhaug SM, Shirk SR, Jensen TK. Therapists' behaviors and youths' therapeutic alliance during trauma-focused cognitive behavioral therapy. J Consult Clin Psychol. 2020 Apr;88(4):350-361. doi: 10.1037/ccp0000465. Epub 2020 Jan 13. PMID 31928035
- [Derived] Lindebo Knutsen M, Sachser C, Holt T, Goldbeck L, Jensen TK. Trajectories and possible predictors of treatment outcome for youth receiving trauma-focused cognitive behavioral therapy. Psychol Trauma. 2020 May;12(4):336-346. doi: 10.1037/tra0000482. Epub 2019 Jul 25. PMID 31343205
- [Derived] Knutsen ML, Czajkowski NO, Ormhaug SM. Changes in posttraumatic stress symptoms, cognitions, and depression during treatment of traumatized youth. Behav Res Ther. 2018 Dec;111:119-126. doi: 10.1016/j.brat.2018.10.010. Epub 2018 Oct 27. PMID 30408700
- [Derived] Aas E, Iversen T, Holt T, Ormhaug SM, Jensen TK. Cost-Effectiveness Analysis of Trauma-Focused Cognitive Behavioral Therapy: A Randomized Control Trial among Norwegian Youth. J Clin Child Adolesc Psychol. 2019;48(sup1):S298-S311. doi: 10.1080/15374416.2018.1463535. Epub 2018 Jun 7. PMID 29877724
- [Derived] Jensen TK, Holt T, Morup Ormhaug S, Fjermestad KW, Wentzel-Larsen T. Change in post-traumatic cognitions mediates treatment effects for traumatized youth-A randomized controlled trial. J Couns Psychol. 2018 Mar;65(2):166-177. doi: 10.1037/cou0000258. PMID 29543473